CLINICAL TRIAL: NCT02676505
Title: Effect of the Length of Second Stage of Labor in Primigravidae on Maternal & Neonatal Outcomes
Acronym: RCT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed El-Sharkawy, Lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Other Study IDs: KasrELAini maternity hospital
Record Dates: First submitted 2015-11-20; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: The Length of Second Labor Stage in Primigravidae on Maternal & Neonatal Outcomes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Group (I)(Coached group):
  It includes 217 patients who are admitted in active stage of labor (cervical dilatation 4cm at least) to labor delivery ward. They are coached by the nurse to use closed-glottis and pushing three to four times during each contraction immediately when cervical dilation reached 10 cm and to continue pushing using this method with each contraction until birth. The nurse counts to 10 during each pushing effort to assist the woman in holding her breath for at least 10 seconds.
  Interventions: Behavioral: Coached pushing group
- 2: It includes 217 patients who are admitted early in active stage of labor (cervical dilatation 4cm at least) to labor delivery ward at 10-cm cervical dilation where they remain until they feel the urge to push or the second stage had lasted 2 hours (whichever came first)., they are encouraged to bear down with contractions without holding their breath (open-glottis) for no more than 6-8 seconds and continue bearing down no more than three times with each contraction until birth.
  Interventions: Behavioral: uncoached pushing group

INTERVENTIONS:
Behavioral: Coached pushing group — It includes 217 patients who are admitted in active stage of labor (cervical dilatation 4cm at least) to labor delivery ward. They are coached by the nurse to use closed-glottis and pushing three to four times during each contraction immediately when cervical dilation reached 10 cm and to continue pushing using this method with each contraction until birth. The nurse counts to 10 during each pushing effort to assist the woman in holding her breath for at least 10 seconds.
  Groups: 1
Behavioral: uncoached pushing group — It includes 217 patients who are admitted early in active stage of labor (cervical dilatation 4cm at least) to labor delivery ward at 10-cm cervical dilation where they remain until they feel the urge to push or the second stage had lasted 2 hours (whichever came first)., they are encouraged to bear down with contractions without holding their breath (open-glottis) for no more than 6-8 seconds and continue bearing down no more than three times with each contraction until birth. .
  Groups: 2

SUMMARY:
The primary purpose of this study is to compare the effects of two different methods of care during the second stage of labor for nulliparous women (coached versus uncoached pushing) on the length of the second stage and how this may affect maternal and neonatal outcome.

DETAILED DESCRIPTION:
The study was conducted on 434 primigravidae women admitted to Kasr El Ainy teaching Maternity Hospital for labor. The study will be done in the period between October 2015 and April 2016. The study will include 434 women with the diagnosis of the first stage of labor with at least cervical dilatation 4cm.

Ethical approval obtained and an informed consent will be taken from each patient after explaining the nature and scope of the study.

Methodology in details:

1. Careful and detailed history taking regarding:

   * Personal history
   * Complaint.
   * History of present pregnancy.
   * Menstrual History.
   * Past history.
2. Careful general examination.
3. Abdominal examination.
4. Local vaginal examination.
5. Ultrasound examination.

Management of Cases:

Group (I)(Coached group):

It includes 217 patients who are admitted in active stage of labor (cervical dilatation 4cm at least) to labor delivery ward. They are coached by the nurse to use closed-glottis and pushing three to four times during each contraction immediately when cervical dilation reached 10 cm and to continue pushing using this method with each contraction until birth. The nurse counts to 10 during each pushing effort to assist the woman in holding her breath for at least 10 seconds.

Group (II)(Uncoached group):

It includes 217 patients who are admitted early in active stage of labor (cervical dilatation 4cm at least) to labor delivery ward at 10-cm cervical dilation where they remain until they feel the urge to push or the second stage had lasted 2 hours (whichever came first)., they are encouraged to bear down with contractions without holding their breath (open-glottis) for no more than 6-8 seconds and continue bearing down no more than three times with each contraction until birth. .

Patients admitted early in labor are subjected to active management of labor as follows:

Pelvic examination performed. Routine amniotomy performed and progress assessed. When dilatation is not increasing, a low dose protocol of oxytocin infusion will be started. Oxytocin diluted in the form of 5IU in 500 ml Ringer lactate making a concentration of nearly 1mu oxytocin/1ml Ringer solution. Infusion instituted at a rate of 1 -2 milliunit (15-30 drops) per minute and increased gradually in increments of 1 -2 milliunit per minute at 30 minutes interval, until at least three uterine contractions noted in a 10 minute period using cardio tocograph.

Assessment of each stage of labor was performed as follow:

1. First stage of labor:

   It includes:
   * Duration of the first stage of labor.
   * Rate of cervical dilatation and foetal descent.
   * Adequacy of uterine contractions and documentation of labor dystocia.
   * Excess uterine activity consisted of uterine tachysystole, hypertonus or uterine hyperstimulation
2. Second stage of labor:

   It includes:
   * Duration of the second stage.
   * Rate of the descent of foetus.
   * Monitoring of foetal heart rate every 5 minutes by sonicaid or continuous by CTG.
   * Use of mediolateral episiotomy.
   * Intervention will be considered either by instrumental delivery,fundal pressure or by CS If the second stage is prolonged more than 2 hours.
   * Monitoring of maternal oxygen saturation by pulse oximeter.
3. Third stage of labor:

   - Duration of the third stage.
4. Assessment of any vaginal laceration or perineal tears with their repair as well as repair of episiotomy.
5. Assessment of quantity of blood loss and assessment of uterine atony(vital instability,number of soaked pads and hemoglobin drop) .
6. Rate of caesarean section during varying stages of labor.
7. Neonatal assessment:

It includes:

* Foetal sex and body weight.
* APGAR score at 1 and 5 minutes..

ELIGIBILITY:
Inclusion Criteria:

All patients admitted in the first stage of labor with cervical dilatation of 4 cm at least:

1. Women age 18-35 years.
2. 37-41 weeks gestation pregnancy.
3. Singleton pregnancy and vertex presentation.
4. Women have no chronic or pregnancy-induced illnesses.
5. Women are in established, spontaneous labor.

Exclusion Criteria:

1. Malpresentation.
2. Women with previous uterine scar.
3. Multiple pregnancy
4. Ante partum hemorrhage.
5. Cephalopelvic disproportion.
6. Women have chronic illnesses.
7. Women with abnormal antenatal period.
8. Patients with foetal distress
9. Premature rupture of membrane
10. Woman having any contraindication to vaginal delivery.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study was conducted on 434 primigravidae women admitted to Kasr El Ainy teaching Maternity Hospital for labor. The study will be done in the period between October 2015 and April 2016. The study will include 434 women with the diagnosis of the first stage of labor with at least cervical dilatation 4cm.
Sampling Method: Probability Sample
Enrollment: 434 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Duration of the second stage | 0-3 hours

SECONDARY OUTCOMES:
Severe maternal morbidity e.g post partum hemorrhage | intrapartum and 2 hours postpartum.
APGAR score after one and five minutes. | 1-5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kasr El Ainy, hospital, Study Director — kasr el ainy street,cairo,egypt